CLINICAL TRIAL: NCT00418860
Title: The Optimal Duration of Dual Antiplatelet Therapy After Implantation of Endeavor Stent in the Patients With Coronary Artery Disease (DATE Registry)
Brief Title: The Optimal Duration of Dual Antiplatelet Therapy After Implantation of Endeavor Stent
Acronym: DATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: HC Gwon, MD,PhD / Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-09-025
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Stent thrombosis; Zotarolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Aspirin, Clopidogrel

INTERVENTIONS:
Drug: Aspirin, Clopidogrel — Aspirin 100mg qd plus clopidogrel 75mg qd for 3 month after index procedure
  Other Names: plavix

SUMMARY:
The purpose of this study to determine whether the dual antiplatelet therapy (aspirin and clopidogrel) for 3 months after coronary implantation of zotarolimus-eluting stent is safe in terms of death, myocardial infarction, or stent thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically significant de novo coronary artery disease
* Stenting only with Endeavor® stents
* The sum of stent length is less than 60 mm for one lesion. The sum of stent length in multiple lesions does not matter.

Exclusion Criteria:

* Cardiogenic shock
* ST-elevation myocardial infarction within 48 hours of symptom onset
* Prior implantation of drug-eluting stents
* Left ventricular dysfunction (echocardiographic left ventricular ejection fraction < 25%)
* Stenting both branch of bifurcation lesion
* Left main trunk lesion
* Graft vessels
* Patients who have to receive clopidogrel due to other conditions
* Patients who have to receive warfarin, cilostazol or other antiplatelet therapy
* Patient with chronic renal failure (S-Cr > 2.0 mg/dl)
* Hypersensitivity to clopidogrel or aspirin
* Expectant survival less than 1 year
* Women who plan to become pregnant
* Patients with bleeding diathesis (coagulopathy, thrombocytopenia or platelet dysfunction, Gastrointestinal or genitourinary bleeding within the prior 3 months)
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence of definite stent thrombosis by Academic Research Consortium Proposed Standard | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea